CLINICAL TRIAL: NCT06203496
Title: Monitoring of Patients With Diffuse Gliomas Using Circulating miRNAs
Acronym: GliomiR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A01732-43
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-12

CONDITIONS: Glioma, Malignant
Keywords: Glioblastoma; Glioma; Biomarker; Radionecrosis
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tumor sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood sample — Blood sample

SUMMARY:
MicroRNAs are small non-coding RNAs involved in the post-transcriptional regulation of genes and, consequently, of intracellular signalling pathways that govern cellular behaviour (Komatsu et al., 2023). They are widely implicated in oncogenesis, and in particular in mechanisms promoting cell migration, invasion and proliferation (Romano et al., 2021). Several preliminary studies have shown that serum levels of pro-oncogenic microRNAs correlate with tumor rates in gliomas (Jones et al., 2021; Levallet et al., 2022; Morokoff et al., 2020). Morokoff's study showed encouraging but insufficient results on the possibility of using microRNAs to differentiate radionecrosis versus recurrence. These results need to be consolidated prospectively, with homogeneous samples taken from all patients.

The aim of this study is to describe the evolution over time of plasma levels of pro-oncogenic microRNAs, after surgery for grade 4 glioma, in order to assess whether they can be used to identify false-positive recurrences on MRI (radionecrosis).

DETAILED DESCRIPTION:
Diffuse gliomas are the most common primary tumors of the central nervous system, representing around 3,400 cases per year in France (Defossez et al., 2019). Their grade varies from 2 to 4. Whatever the grade, their prognosis is dismal (Grade 2: median survival > 10 years, Grade 3: median survival around 5 years, Grades 4: median survival < 2 years) (Yang et al., 2016).

Grade 4 diffuse gliomas are the most common gliomas. Their treatment is based on excision of the tumor as completely as possible while preserving the patient's neurological functions. This surgical treatment is followed by a "Stupp" radiochemotherapy protocol (Stupp et al., 2005). Nevertheless, recurrence of grade 4 gliomas after surgery is inevitable, and usually occurs within 2 years of surgery (Pineda et al., 2023). In fact, gliomas are infiltrating tumors, with tumor cells infiltrating the brain parenchyma up to 2 cm from the periphery of the tumor visualized on MRI, which explains their inevitable recurrence, since surgery cannot be wide (it is difficult to achieve "safety margins" at the cerebral level) and will invariably leave tumor cells in situ (Pallud et al., 2013).

In the event of recurrence, second-line chemotherapy or further surgery may then be proposed to the patient. Patients are monitored by regular brain MRI scans, but it is important to be aware of the risks involved.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Grade 4 diffuse glioma
* Surgery in the neurosurgery department of Caen University Hospital
* Patient affiliated to a social security scheme
* Patient followed at Caen University Hospital
* No opposition from patient

Exclusion Criteria:

* - Patients who underwent biopsy (lack of material for study, limited interest of monitoring for these patients without surgical excision).
* Patients with grade 1 circumscribed glioma or grade 2 or 3 diffuse glioma.
* Other non-glial histologies, glioneuronal histology
* Minor patients
* Patient not affiliated to a social security scheme
* A minor under guardianship or protection
* Patient opposed to study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with surgically resected grade 4 glioma
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of glioma on MRI | 2 years
  Aspect of recurrence on MRI

SECONDARY OUTCOMES:
OS | 2 years
  Overall Survival
PFS | 2 years
  Progression free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Arthur Leclerc, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levallet G, Dubois F, Leclerc A, Petit E, Bekaert L, Faisant M, Creveuil C, Emery E, Zalcman G, Lechapt-Zalcman E. The Use of Pro-Angiogenic and/or Pro-Hypoxic miRNAs as Tools to Monitor Patients with Diffuse Gliomas. Int J Mol Sci. 2022 May 27;23(11):6042. doi: 10.3390/ijms23116042. PMID 35682718
- [Background] Komatsu S, Kitai H, Suzuki HI. Network Regulation of microRNA Biogenesis and Target Interaction. Cells. 2023 Jan 13;12(2):306. doi: 10.3390/cells12020306. PMID 36672241
- [Background] Morokoff A, Jones J, Nguyen H, Ma C, Lasocki A, Gaillard F, Bennett I, Luwor R, Stylli S, Paradiso L, Koldej R, Paldor I, Molania R, Speed TP, Webb A, Infusini G, Li J, Malpas C, Kalincik T, Drummond K, Siegal T, Kaye AH. Serum microRNA is a biomarker for post-operative monitoring in glioma. J Neurooncol. 2020 Sep;149(3):391-400. doi: 10.1007/s11060-020-03566-w. Epub 2020 Sep 11. PMID 32915353